CLINICAL TRIAL: NCT05914597
Title: 5G SUCCEEDS Trial Feasibility of Home Delivery of Colon Capsule Endoscopy Service With the Help of 5 G Technology
Brief Title: Trial Feasibility of Home Delivery of Colon Capsule Endoscopy Service With the Help of 5 G Technology
Acronym: 5GSUCCEEDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Dr Gohar Jalayeri Nia, Dr Gohar Jalayeri Nia, National Health Service, United Kingdom
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 311685
Record Dates: First submitted 2022-06-30; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Colon Capsule Endoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Assessing the acceptance of remote colon capsule endoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant (Other): Patients with lower gastrointestinal symptoms who have been selected by overseeing clinician meeting NHS England criteria to undergo colon capsule endoscopy as part of their standard of care and are 18 or over .
  Interventions: Other: Setting up home delivery of Colon capsule endoscopy

INTERVENTIONS:
Other: Setting up home delivery of Colon capsule endoscopy — Feasibility study of home delivery of CCE

SUMMARY:
Patients without alarming symptoms are at low risk of bowel cancer . However, in majority of those patients colonoscopy (gold standard) is needed to diagnose colorectal cancer or other non-neoplastic conditions such as Inflammatory bowel disease . Evaluation of patients with lower gastrointestinal symptoms ( low-intermediate risk group) represent significant pressure for colonoscopy services . At the end of August 2019 there were a total 44,388 patients still waiting for colonoscopy.

Covid 19 pandemic has placed significant pressure on healthcare systems since March 2020.The aerosol generating potential of endoscopy has led to multiple Gastroenterology and Endoscopy societies suggesting immediate cessation of all but emergency colonoscopy during the peak phase of the pandemic which put colonoscopy capacity even more under pressure Data from the National Endoscopy Database indicate that total endoscopic activity fell rapidly to 5% of normal levels during the peak phase of the COVID-19 epidemic in the UK (from approximately 35 000 reported procedures per week to 1700, for the week ending 13 April .

In order to reduce potential diagnostic delays as a result of COVID pandemic , the role of colon capsule endoscopy (CCE) as a non invasive diagnostic test is being increasingly recognise, which allows for a pain-free colonic assessment by eliminating the need for instrument insertion, gas insufflation or sedation .

The aim of the 5G SUCCEEDS study is to trial feasibility of home delivery of Colon Capsule Endoscopy service with the help of 5 G technology. Currently patients need to attend hospital to access this service.

DETAILED DESCRIPTION:
According to the European Society of Gastrointestinal Endoscopy (ESGE), CCE can be used in average-risk patients for CRC screening and as an adjunctive test in patients with a prior incomplete Colonoscopy, or in whom the latter is contraindicated or refused CCE. Therefore, it is a potentially beneficial method of investigating patients by reducing the pressure on the restricted endoscopy services in the post-COVID era. In line with that, the NHS England is implementing a pilot project of CCE in patients referred on the two weeks wait pathway. The purpose of this study is to provide an alternative diagnostic test, while colonoscopy investigations are delayed due to the COVID Pandemic. This initially is undertaken in those at low risk of colorectal cancer. Low risk patients will have low levels of blood in the stool measured by FIT. Those at high risk will proceed straight to colonoscopy .

At present in order to perform the CCE procedure it still requires patients to attend hospital, usually carried out by one healthcare professional. It involves ﬁtting a receiver belt to the patient and oral administration of the disposable capsule. Therefore we propose a different mode of delivery to avoid hospital visit in order to mitigate COVID risk, in line with integrated care system of delivery away from hospital.

We believe implementing digitally-enabled care will significantly reduce travel and journeys to hospital and will contribute to care closer to home. Setting up CCE home delivery system can facilitate many sustainability benefits including reduction or repurposing of estate footprint, reduced local air pollution, increased patient wellbeing /choice and time savings for the workforce . By implying new digital technology such as 5G we will be able to deliver the CCE service more effectively and productively, with patients at the centre which is in line with NHS X digital strategy .

The aim of this study is to trial feasibility of home delivery of Colon Capsule Endoscopy service with the help of 5 G technology. Currently patients need to attend hospital to access this service.

The term "5G" refers to the fifth generation of wireless transmission technology, expected to have a significant influence in many aspects of contemporary society, including healthcare. Based on 5G super bandwidth per unit area, connectivity, coverage (up to 100%), and capacity to connect devices per unit will lead to an ecosystem in which an "intelligence network" can serve real-time interactivity for massive medical equipment and patients' wearable devices, with cloud computing-based trade-offs between speed, latency, coverage, availability. COVID-19 has caused widespread healthcare impact .Countries and healthcare systems around the world have been forced to rapidly adapt to tele-health and digital innovations to mitigate the impact of the risk of virus transmission to what is widely regarded as the "new normal". With 5G technology, which has lower latency and higher capacity, healthcare systems can provide the care their patients need and expect remotely .

Working with specialist connectivity partners, the CCE smartbox has been developed by CorporateHealth International, an Inverness-based capsule endoscopy service provider. A device supported by 5 G can be used independently in patient's homes. The Smartbox will be utilised to make telecommunication with the patient robust and safe, reducing the risk of failed procedure attempts. Faster and reliable 5G internet will enable the use of a 'virtual assistant' that can provide answers and guidance to the patient while clinicians can track and monitor the location of the equipment throughout the process. It is anticipated that the adoption of 5G to enable home testing will reduce waiting times and speed up the process of identifying irregularities and any subsequent treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been selected by overseeing clinician meeting NHS England criteria to undergo colon capsule endoscopy as part of their standard of care
* Age between 18-55

Exclusion Criteria:

* Patients unable or unwilling to provide consent to take part in the study
* Patient is pregnant
* Standard CCE exclusion criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of home delivery of CCE service | 12month
  To assess the feasibility of Colon Capsule Endoscopy home delivery service, we followed a structured approach. We are aiming to deliver the whole CCE service at home by using a smartbox, 5G technology and telemedicine communication to conduct the study and troubleshoot any upcoming issues. The target population is based on the number of available smartboxes. Through a comprehensive process we obtained all the regulatory and ethical approval for conducting the study

SECONDARY OUTCOMES:
assessing the patient's acceptability of home delivery of CCE service | 6 month
  One of the main aims of this study is to measure the patient' satisfaction. We design the questionnaire to capture the necessary information. We wanted to include factors such as quality of care, experience with using the capsule endoscopy equipment and smartbox at home, and overall experience. Format of the questionnaire is mainly structured with closed-ended questions (multiple-choice or Likert scale. When we are using a scale from 0 to 5, 0 represents extremely easy and 5 represents extremely difficult. Based on our identified domains, we develop specific questions that assess patient satisfaction within each domain, and we ensure that the questions are clear, concise, and unambiguous and we avoided leading or biased questions that may influence the responses.

CONTACTS AND LOCATIONS:
Overall Officials: Gohar J Nia, MD, Principal Investigator — National Health System United Kingdom; Professor Ramesh Arasaradnam, PHD, Study Director — National Health System United Kingdom
Locations (1):
- Gohar jalayeri Nia, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We are aiming to share IPD to other researchers such as protocol and CSR
Supporting Information: Study Protocol, CSR
Time Frame: 12 month